CLINICAL TRIAL: NCT04410367
Title: An Open-label, Single-arm, Single-dose, Prospective, Multicenter Phase 2b Study to Establish Image Interpretation Criteria for 18F-Fluciclovine Positron Emission Tomography (PET) in Detecting Recurrent Brain Metastases After Radiation Therapy
Brief Title: Study to Establish Image Interpretation Criteria for 18F Fluciclovine PET in Detecting Recurrent Brain Metastases (PURSUE)
Acronym: PURSUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Precision For Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-FLC-219
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Brain Metastases
Keywords: Recurrent Brain Metastases; Diagnostic; Positron Emission Tomography (PET) Scan
MeSH Terms: conditions — Brain Neoplasms; Disease | interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Positron Emission Tomography (PET) Imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Single intravenous administration of 18F fluciclovine for PET Scan
  Interventions: Drug: 18F fluciclovine

INTERVENTIONS:
Drug: 18F fluciclovine — 18F fluciclovine injection, 185 MegaBecquerel (MBq) (5 Millicurie (mCi)) ± 20%, delivered as an intravenous bolus
  Other Names: Axumin

SUMMARY:
An Open-label, Single-arm, Single-dose, Prospective, Multicenter Phase 2b Study to Establish Image Interpretation Criteria for 18F-Fluciclovine Positron Emission Tomography (PET) in Detecting Recurrent Brain Metastases After Radiation Therapy

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
2. Previous history of solid tumor brain metastasis of any origin
3. Histopathological confirmation of the primary solid tumor or a metastatic site
4. Previous radiation therapy of brain metastatic lesion(s)
5. A reference lesion considered by the site investigator to be equivocal for recurrent brain metastasis
6. Patient requires further confirmatory diagnostic procedures to confirm brain MRI findings and is planned for craniotomy

Exclusion Criteria:

1. Patients with a history of active hematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Teoh, MD, Study Director — Blue Earth Diagnostics; Rupesh Kotecha, MD, Principal Investigator — Miami Cancer Institute
Locations (9):
- United States (9):
  - John Wayne Cancer Institute at Providence St. John's Health Center, Santa Monica, California
  - Yale School of Medicine, New Haven, Connecticut
  - Miami Cancer Institute, Miami, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University School of Medicine Center for Clinical Imaging Research, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - University Hospital Cleveland, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Center for Quantitative Cancer Imaging at Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a history of brain metastases previously treated with primary, adjuvant, or repeat (salvage) radiation therapy, with a recent standard of care (SoC) brain magnetic resonance imaging (MRI) found to be equivocal for recurrent brain metastasis, and who met all the inclusion criteria and none of the exclusion criteria, were consented and enrolled.
  Subjects were screened between 28Oct2020 and 30Dec2021. Nine clinical research sites in the US participated in the study.
Pre-assignment Details: On-study site investigators prospectively annotated and measured the 'reference lesion' on a postradiation treatment MRI scan and on the SoC MRI brain scan to confirm eligibility. The 'reference lesion' was defined as the lesion which was Equivocal for recurrent metastasis on SoC MRI, Intended for pre-planned SoC craniotomy, and If > 1 equivocal lesion was intended for resection, the largest of these lesions.
Groups:
- 18F-Fluciclovine Injection: Subjects who have been dosed with 18F-Fluciclovine, have an evaluable on-study PET scan, and an evaluable central histopathology report from the sample obtained from the SoC craniotomy.
Period: Overall Study
Arm/Group | 18F-Fluciclovine Injection
Started | 23
Underwent 18F-fluciclovine PET | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients: Single intravenous administration of 18F fluciclovine for PET Scan
  18F fluciclovine: 18F fluciclovine injection, 185 MBq (5 mCi) ± 20%, delivered as an intravenous bolus
Arm/Group | Patients
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of 18F Fluciclovine PET for Detecting Recurrent Brain Metastases at Different Visual Thresholds
Description: Sensitivity is calculated as % of participants with positive histopathology who are classified as positive on their 18F fluciclovine PET (i.e. true positive). Each participant had one lesion, therefore results are representative of both subject and lesion level sensitivity.
  Three readers evaluated the PET scans to classify 18F fluciclovine uptake in study lesions according to 4 incremental categories: absent, mild, moderate or marked. Three different thresholds of 18F fluciclovine uptake were then applied to calculate the sensitivity: Mild or Higher Uptake, Moderate or Higher Uptake, Marked Uptake. As an example, for calculating sensitivity based on the threshold of Mild or Higher Uptake, all participants with positive histopathology, classified by a reader as having mild, moderate or marked 18F fluciclovine uptake, would be categorized as true positive. This calculation was then repeated on the other two threshold categories, to produce sensitivities at different thresholds.
Time Frame: 60 days
Population: Sensitivity analysis (%) based on 10 subjects with positive lesions per standard of truth (central histopathological analysis).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 18F-Fluciclovine Injection: Subjects who have been dosed with 18F-Fluciclovine, have an evaluable on-study PET scan, and positive histopathology.
Arm/Group | 18F-Fluciclovine Injection
Number analyzed (Participants) | 10
percentage of participants
  Mild or Higher Uptake = Positive : Central Reader 1 | 100 [69.2 to 100]
  Mild or Higher Uptake = Positive : Central Reader 2 | 100 [69.2 to 100]
  Mild or Higher Uptake = Positive : Central Reader 3 | 100 [69.2 to 100]
  Moderate or Higher Uptake = Positive : Central Reader 1 | 100 [69.2 to 100]
  Moderate or Higher Uptake = Positive : Central Reader 2 | 100 [69.2 to 100]
  Moderate or Higher Uptake = Positive : Central Reader 3 | 90 [55.5 to 99.8]
  Marked Uptake = Positive : Central Reader 1 | 80 [44.4 to 97.5]
  Marked Uptake = Positive : Central Reader 2 | 40 [12.2 to 73.8]
  Marked Uptake = Positive : Central Reader 3 | 60 [26.2 to 87.8]

2. Primary Outcome: Specificity of 18F Fluciclovine PET for Detecting Recurrent Brain Metastases at Different Visual Thresholds
Description: Specificity is calculated as the % of participants with negative histopathology who are classified as negative on their 18F fluciclovine PET (i.e. true negative). Each participant had 1 lesion, therefore results are representative of both subject and lesion level specificity. 3 readers evaluated the PET scans to classify 18F fluciclovine uptake in study lesions according to 4 incremental categories: absent, mild, moderate or marked. 3 different thresholds of uptake were then applied to calculate the specificity: Mild or Higher Uptake, Moderate or Higher Uptake, Marked Uptake. Example, for calculating specificity based on the threshold of Moderate or Higher Uptake, all participants with negative histopath, classified by a reader as having absent or mild uptake (i.e. not classified by a reader as having moderate or marked uptake), would be categorized as true negative. This calculation was repeated on the other 2 threshold categories, to produce specificities at different thresholds
Time Frame: 60 days
Population: Specificity analysis (%) based on 13 subjects with negative lesions per standard of truth (central histopathological analysis).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 18F-Fluciclovine Injection: Subjects who have been dosed with 18F-Fluciclovine, have an evaluable on-study PET scan, and negative histopathology.
Arm/Group | 18F-Fluciclovine Injection
Number analyzed (Participants) | 13
percentage of participants
  Mild or Higher Uptake = Positive : Central Reader 1 | 0 [0.0 to 24.7]
  Mild or Higher Uptake = Positive : Central Reader 2 | 0 [0.0 to 24.7]
  Mild or Higher Uptake = Positive : Central Reader 3 | 0 [0.0 to 24.7]
  Moderate or Higher Uptake = Positive : Central Reader 1 | 38.5 [13.9 to 68.4]
  Moderate or Higher Uptake = Positive : Central Reader 2 | 30.8 [9.1 to 61.4]
  Moderate or Higher Uptake = Positive : Central Reader 3 | 46.2 [19.2 to 74.9]
  Marked Uptake = Positive : Central Reader 1 | 92.3 [64.0 to 99.8]
  Marked Uptake = Positive : Central Reader 2 | 100 [75.3 to 100.0]
  Marked Uptake = Positive : Central Reader 3 | 100 [75.3 to 100.0]

3. Secondary Outcome: Sensitivity of 18F Fluciclovine PET for Detecting Recurrent Brain Metastases Based on Quantitative and Dynamic Measures of Lesion 18F Fluciclovine Uptake
Description: Sensitivity calculated as %participants with positive histopath and positive on PET (i.e. true positive). Each participant had 1 lesion, results represent both subject and lesion level sensitivity. Sensitivity is calculated using positive PET classified by quantitative and dynamic measures. Quantitative measure is based on lesion standardized uptake value (SUV). Receiver Operating Characteristic (ROC) analysis of all participant lesion SUV was performed. ROC analyses was performed to select a SUV threshold for calculating sensitivity. Sensitivity calculation: participants with positive histopath and SUV = or > threshold are positive on scan. Dynamic measure: 3 readers evaluated PET scans to classify uptake pattern based on 4 categories: Type 0, Type I, Type II, Type III. Sensitivity is calculated for each type of uptake pattern (example: calculating sensitivity based on Type I pattern, participants with positive histopath, classified as Type I, would be categorized as true positive).
Time Frame: 60 days
Population: Sensitivity analysis (%) based on 10 subjects with positive lesions per standard of truth.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 18F-Fluciclovine Injection
Number analyzed (Participants) | 10
percentage of participants
  Quantitative SUV ≥ 4.8 = Positive : Central Reader 1 | 80 [44.4 to 97.5]
  Quantitative SUV ≥ 4.8 = Positive : Central Reader 2 | 80 [44.4 to 97.5]
  Quantitative SUV ≥ 4.8 = Positive : Central Reader 3 | 80 [44.4 to 97.5]
  Dynamic Type 0: Central Reader 1 | 0 [0 to 30.9]
  Dynamic Type 0 : Central Reader 2 | 0 [0 to 30.9]
  Dynamic Type 0 : Central Reader 3 | 0 [0 to 30.9]
  Dynamic Type I: Central Reader 1 | 80 [44.4 to 97.5]
  Dynamic Type I: Central Reader 2 | 90 [55.5 to 99.8]
  Dynamic Type I: Central Reader 3 | 100 [69.2 to 100]
  Dynamic Type II: Central Reader 1 | 10 [0.3 to 44.5]
  Dynamic Type II: Central Reader 2 | 10 [0.3 to 44.5]
  Dynamic Type II: Central Reader 3 | 0 [0 to 30.9]
  Dynamic Type III: Central Reader 1 | 10 [0.3 to 44.5]
  Dynamic Type III: Central Reader 2 | 0 [0 to 30.9]
  Dynamic Type III: Central Reader 3 | 0 [0 to 30.9]

4. Secondary Outcome: Specificity of Different Thresholds of Quantitative and Dynamic Measures of Lesion 18F Fluciclovine Uptake.
Description: Specificity is calculated as %participants with negative histopath and negative on PET (i.e. true negative). Each participant had 1 lesion, results represent both subject and lesion level specificity. Specificity is calculated using negative PET classified by quantitative and dynamic measures. Quantitative measure is based on lesion standardized uptake value (SUV). Receiver Operating Characteristic (ROC) analysis of all participant lesion SUV was performed. ROC analyses was performed to select a SUV threshold for calculating sensitivity. Specificity calculation: participants with negative histopath, SUV < threshold are negative on scan. Dynamic measure: 3 readers evaluated PET scans to classify uptake pattern based on 4 categories: Type 0, Type I, Type II, Type III. Specificity is calculated for each type of uptake pattern (example, calculating specificity based on Type I pattern, participants with negative histopath, classified as Type I, would be categorized as true negative)
Time Frame: 60 days
Population: Subjects who have been dosed with 18F-Fluciclovine, have an evaluable on-study PET scan, and negative histopathology.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 18F-Fluciclovine Injection: Specificity of 18F fluciclovine PET for detecting recurrent brain metastases based on quantitative and dynamic measures of lesion 18F fluciclovine uptake
Arm/Group | 18F-Fluciclovine Injection
Number analyzed (Participants) | 13
percentage of participants
  SUV ≥ 4.8 : Central Reader 1 | 84.6 [54.6 to 98.1]
  SUV ≥ 4.8 : Central Reader 2 | 84.6 [54.6 to 98.1]
  SUV ≥ 4.8 : Central Reader 3 | 84.6 [54.6 to 98.1]
  Dynamic Type 0 : Central Reader 1 | 100 [75.3 to 100]
  Dynamic Type 0 : Central Reader 2 | 100 [75.3 to 100]
  Dynamic Type 0 : Central Reader 3 | 100 [75.3 to 100]
  Dynamic Type I : Central Reader 1 | 7.7 [0.2 to 36.0]
  Dynamic Type I : Central Reader 2 | 15.4 [1.9 to 45.5]
  Dynamic Type I : Central Reader 3 | 0 [0 to 24.7]
  Dynamic Type II : Central Reader 1 | 92.3 [64.0 to 99.8]
  Dynamic Type II : Central Reader 2 | 84.6 [54.6 to 98.1]
  Dynamic Type II : Central Reader 3 | 100 [75.3 to 100]
  Dynamic Type III : Central Reader 1 | 100 [75.3 to 100]
  Dynamic Type III : Central Reader 2 | 100 [75.3 to 100]
  Dynamic Type III : Central Reader 3 | 100 [75.3 to 100]

5. Secondary Outcome: Treatment-emergent Adverse Events
Description: Safety will be assessed from data on the occurrence of one or more treatment-emergent Adverse Events from the time of intravenous administration of 18F fluciclovine until 1 day post-18F-fluciclovine administration.
Time Frame: From the time of administration of 18F fluciclovine until 1 day post-18F-fluciclovine administration.
Measure: Count of Participants; unit: Participants
Groups:
- 18F-Fluciclovine Injection: Safety will be assessed from data on the occurrence of one or more treatment-emergent Adverse Events from the time of intravenous administration of 18F fluciclovine until 2 days post-18F-fluciclovine administration.
Arm/Group | 18F-Fluciclovine Injection
Number analyzed (Participants) | 23
Participants
  Subjects reporting at least 1 TEAE | 1
  Nervous System Disorders (Headache) | 1

ADVERSE EVENTS:
Time Frame: Safety was assessed from the time of 18F-fluciclovine administration until 1 day post18Ffluciclovine administration based on reported adverse events (AEs) and serious adverse events (SAEs); treatment emergent adverse events (TEAE).
Arm/Group | 18F-Fluciclovine Injection
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-Fluciclovine Injection (N=23)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the INSTITUTION nor the INVESTIGATOR will submit for publication or public disclosure any publication or disclosure based on the results of the Study until after the first to occur of (a) publication of the multi-center clinical trial results; (b) notification by BED that the multi-center clinical trial submission is no longer planned; or (c) the eighteen (18) month anniversary of the completion or early termination of the multi-center clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04410367/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04410367/SAP_003.pdf